CLINICAL TRIAL: NCT04005079
Title: A Prospective Randomized Control Trial of Pilocarpine Use After Combined Cataract/Trabectome Surgery
Brief Title: Pilocarpine After Combined Cataract/Trabectome Surgery
Acronym: PACCT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: not performing Trabectomes
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8704
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Cataract surgery; Trabectome; Eye Surgery; Vision; Glaucoma Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Pilocarpine; Ofloxacin; Prednisolone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: The "Treatment Group" will use 2% pilocarpine in the postoperative period in addition to standard post-operative drops (Prednisolone acetate and Ofloxacin). The "Control Group" will use only Prednisolone acetate and Ofloxacin, without pilocarpine.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): 2% pilocarpine and standard of care post op drops ( Prednisolone acetate and Ofloxacin)
  Interventions: Drug: Pilocarpine; Drug: Ofloxacin; Drug: Prednisolone
- Control Group (Active Comparator): Standard of care post op drops-Prednisolone acetate and Ofloxacin, without pilocarpine
  Interventions: Drug: Ofloxacin; Drug: Prednisolone

INTERVENTIONS:
Drug: Pilocarpine — 2% pilocarpine in the postoperative period in addition to standard postoperative drops (Prednisolone acetate and Ofloxacin)
  Other Names: Ocu-Carpine
  Arms: Treatment Group
Drug: Ofloxacin — Standard of care
  Other Names: Ocuflox
Drug: Prednisolone — Standard of Care
  Other Names: Ocu-Pred

SUMMARY:
Combined cataract + trabectome surgery is a surgery designed to help lower the intraocular pressure (pressure in the eye) and hopefully reduce the need for topical drops, progression of glaucoma, and/or further glaucoma surgeries. The purpose of this study is to assess whether using pilocarpine, a medication which is FDA approved to induce miosis, (in other words cause the pupil to constrict or become smaller) provides additional benefit to the success of Trabectome and cataract surgery.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, and its treatment consists of lowering intraocular pressure (IOP) to prevent damage to the optic nerve and loss of vision. Microincisional glaucoma surgery (MIGS) have become more popular in recent years as less invasive methods than traditional surgeries that effectively reduce IOP and help reduce the medication burden on patients.There are multiple available MIGS procedures, most of which act by increasing trabecular outflow. One such procedure is the Trabectome, which is usually performed in combination with cataract surgery.

Trabectome is an FDA approved device used to perform a trabeculectomy via an internal approach. A strip of 60-120 degrees of the nasal angle trabecular meshwork and the inner wall of Schlemm's canal are removed providing a direct pathway for aqueous outflow from the anterior chamber into the collector channels[2].

Pilocarpine, a parasympathomimetic agent, is a glaucoma medication that works by causing contraction of the ciliary muscle leading to opening of the trabecular meshwork[3]. Due to its frequent dosing requirement and large number of ocular and systemic side effects, pilocarpine has largely fallen out of favor for the treatment of primary open angle glaucoma (POAG), except in patients for whom few other alternatives exist. However, pilocarpine is often used after trabectome surgery.

The rationale for its use after Trabectome procedure is for its miotic effect, which theoretically may prevent the formation of peripheral anterior synechiae. Formation of peripheral anterior synechiae can lead to the closure of the cleft that is generated and the possibility of failure of the procedure. While the theoretical benefit of pilocarpine has been proposed, its actual benefit has never been proven.

In this study, the aim is to evaluate whether Trabecome / Cataract surgery without pilocarpine is non-inferior to Trabecome / Cataract surgery procedure followed by treatment with pilocarpine

ELIGIBILITY:
Inclusion Criteria:

* Age Range: 30 to 100 years old
* Patients with ocular hypertension or open angle glaucoma undergoing combined cataract surgery with trabectome in a single surgical center

Exclusion Criteria:

* Patients with previous history of eye surgeries (including laser procedures).

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Percentage of intraocular lowering from baseline | Up to 1 year
  Percentage of IOP drop at 1 month, 6 months and 1 year after surgery.
Number of IOP lowering agents required to achieve goal IOP | Up to 3 years
  The number of pre and post procedure drops required to achieve goal IOP at 6 months, 1, 2 and 3 years after combined cataract/trabectome surgery in patients treated with post-op pilocarpine vs control
Rate of progression to further glaucoma surgeries. | Up to 3 years
  Assessment of the rate of progression towards further surgery in patients treated with post-op pilocarpine vs control over a 3 year follow up period

SECONDARY OUTCOMES:
Frequency of pilocarpine related side effects | Up to 3 years
  Most common side effects will be counted - blurry vision, decrease night vision, headaches, browache, nausea, vomiting, diarrhea
Frequency of drug discontinuation due to pilocarpine related side effects | Up to 3 years
  The number of drug discontinuation due to common side effects will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jeng (Melissa) Yao, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04005079/Prot_SAP_000.pdf